CLINICAL TRIAL: NCT04778436
Title: Macular Drusen Evolution in Patients With Intermediate Age-related Macular Degeneration (AMD) Taking Oral Food Supplementation: an Open-label,Single-arm Pilot Study
Brief Title: Macula Evolution in Patients With AMD Taking Oral Food Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LT7082-001
Record Dates: First submitted 2021-01-18; First posted 2021-03-03 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: an open-label, single-arm, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T7082 (Experimental): After inclusion, the patients will consume an association of 4 food supplements including Nutrof Total.
  Interventions: Dietary Supplement: T7082

INTERVENTIONS:
Dietary Supplement: T7082 — Patients will take food supplementation for 12 months. For each patient : 5 visits with ophthalmogist and 6 phone call

SUMMARY:
LT7082-001 is an open-label, single-arm pilot study. Patients with intermediate age-related macular degeneration (AMD) wil take T7082 during 12 months , an association of 4 food supplementations .

The study objectives are to describe morphological changes and evolution of drusen in macula after a 12-month of food supplementation and to assess the safety of T7082

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated
* Age ≥ 50 years old
* At least one Eligible Eye, defined by following conditions :

  1. Far Best Corrected Visual Acuity (BCVA) ≥ 75 ETDRS letters (or ≥ 20/32 Snellen equivalent)
  2. At least one drusen with a minimal diameter of 125 µM assessed by SD-OCT / intermediate age-related macular degeneration
  3. Macula sparing
  4. Clear ocular media
  5. Adequate pupillary dilation

Exclusion Criteria:

* Presence of other macular disease such as epiretinal membrane or macular telangiectasia.
* Presence of any geographic atrophy including macular region
* Any history of retina neovascularization
* Macula or retinal diseases other than age-related macular degeneration
* A concurrent ocular pathology that may contribute to vision loss (eg, choroidal neovascularization, glaucoma, visually significant cataract, optic neuropathy, history of retinal surgery) or interfere with acquisition of high-quality images
* Ocular or periocular infections
* Presence of congenital retinal pathologies that may impact data collection
* Exudative AMD

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
evolution of drusen in the macula | 2 months, 5 months 8 months and 12 months
  Change from baseline in drusen region in 4 categories (disappearance, decrease, stable, increase) at 2, 5 and 6 months by Optical Coherence Tomography (OCT-SD)
morphological changes in the macula | 2 months, 5 months 8 months and 12 months
  Presence and/or evolution of atrophic area (Yes/No) at 2, 5, 6 and 12 months assessed by autofluorescence
Treatment-Emergent Adverse events (TEAE), Serious treatment-emergent adverse events (STEAE), Treatment-Emergent Adverse Reaction (TEAR) | 2 months, 5 months 8 months and 12 months
  Frequency of TEAE,STEAE,TEAR

CONTACTS AND LOCATIONS:
Locations (1):
- Wilfried Roquet, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No